CLINICAL TRIAL: NCT03765710
Title: Role of Dietary Protein Intake on Whole Body Protein Balance in Elderly Adults
Brief Title: Role of Dietary Protein Intake in Elderly Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 204291
Record Dates: First submitted 2018-11-26; First posted 2018-12-05 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2018-12

CONDITIONS: Protein Overload

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recommended protein intake (Experimental): Subjects consumed a mixed meal with a macronutrient distribution of 13% protein, 54% carbohydrate, and 33% fat.
  Interventions: Other: Recommended protein intake
- Elevated protein intake (Experimental): Subjects consumed a mixed meal with a macronutrient distribution of 26% protein, 44% carbohydrate, and 30% fat.
  Interventions: Other: Elevated protein intake

INTERVENTIONS:
Other: Recommended protein intake — Recommended protein intake in a mixed meal contained 13% protein, 54% carbohydrate, and 33% fat.
  Arms: Recommended protein intake
Other: Elevated protein intake — Increased protein intake in a mixed meal contained 26% protein, 44% carbohydrate, and 30% fat.
  Arms: Elevated protein intake

SUMMARY:
The investigators examined the effects of dietary protein intake in a mixed meal at two levels of protein amount on whole body protein metabolisms in older adults.

DETAILED DESCRIPTION:
The investigators determined the total anabolic response to an amount of protein intake commonly eaten with dinner (70g) as compared with the amount required to maximally stimulate muscle protein synthesis (35g). Men and women, ages > 60 years will be studied under two levels of protein intake in mixed meals in random order (35g or 70g protein in isocaloric mixed meals). For two days prior to each stable isotope tracer study, subjects' dietary intake of calories and protein will be stabilized by providing subjects their entire diets. On the third day, a 8-hr metabolic study will be conducted in the UAMS Reynolds Institute on Aging (IOA) to determine the total anabolic response to the particular amount of beef intake, which will be repeated with the other amount of protein in mixed meal after a minimum 7-day washout interval. The investigators measured whole body protein kinetics, muscle fractional synthetic rate, and plasma amino acid profile.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, ages > 60 years

Exclusion Criteria:

* History of diabetes
* History of malignancy in the 6 months prior to enrollment
* History of gastrointestinal bypass surgery (Lapband, etc)
* History of a chronic inflammatory condition or disease (Lupus, HIV/AIDS, etc)
* Pregnant females
* Subjects who do not or will not eat animal proteins
* Subjects who cannot refrain from consuming protein or amino acid supplements during their participation in this study
* Subjects who report regular resistance exercise (more than once per week)
* Hemoglobin less than 9.5 mg/dL at the screening visit
* Platelets less than 150,000 at the screening visit
* Subjects who are not willing or able to suspend aspirin for several days prior to their muscle biopsies
* Subjects who have been prescribed a blood-thinning medication (Coumadin, lovenox, heparin, Plavix, etc.)
* Concomitant use of corticosteroids (ingestion, injection or transdermal)
* Any other disease or condition that would place the subject at increased risk of harm if they were to participate, at the discretion of the study physician

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Changes in whole body anabolism | Change before and after a mixed meal intake for approximately 8 hours
  Whole body net protein balance in gram protein
Changes in skeletal muscle synthetic rate | Change before and after a mixed meal intake for approximately 8 hours
  Skeletal muscle fractional synthetic rate in % synthesis